CLINICAL TRIAL: NCT06809686
Title: An Observational Study to Collect High Resolution 12-Lead Electrocardiogram (ECG) Data for the Development of an ECG Library to Support the Development of a Tool to Monitor Disease Progression, Gather Patient Perspectives on Standard of Care Heart Failure Procedures and Facilitate Familiarity with the Clinical Trial Environment in Patients with Heart Failure with Mildly Reduced or Preserved Ejection Fraction
Brief Title: Study to Collect High-Resolution ECG Data and Patient Insights on Heart Failure Care
Status: Recruiting | Type: Observational
Sponsor: Richmond Research Institute (Industry)
Responsible Party: Sponsor
Organization: Richmond Pharmacology Limited (Industry)
Other Study IDs: C24042
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Haematology, coagulation, biochemistry Serology (HIV 1 and 2, Hepatitis B & C) COVID-19 and Influenza test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Heart Failure with Mildly Reduced or Preserved Ejection Fraction: Study to Collect High Resolution 12-Lead Electrocardiogram (ECG) Data for the Development of an ECG Library to Support the Development of a Tool to Monitor Disease Progression, Gather Patient Perspectives on Standard of Care Heart Failure Procedures and Facilitate Familiarity with the Clinical Trial Environment in Patients with Heart Failure with Mildly Reduced or Preserved Ejection Fraction

SUMMARY:
The purpose of this study is to establish an electrocardiogram (ECG) data library to facilitate future studies on heart disease. Additionally, the study will be used to monitor changes in the patient's standard of care throughout the study period and gather patient perspectives on routine diagnostic procedures and disease monitoring and feedback on the design of heart failure trials.

DETAILED DESCRIPTION:
Patients with heart failure with mildly reduced or preserved ejection fraction will be invited to participate in this patient observational study.

After providing informed consent, participants will then undergo a series of clinical assessments, and the participants' ECGs will be used to contribute to establishing an ECG library for future heart disease research. Additionally, patients' perspectives on the current standard of care clinical procedures will be gathered. Patient preferences will be gathered in relation to factors around routine clinical investigations for heart failure to better design a disease monitoring tool to include clinical and patient preferences. Also, the patients may be updated on the latest therapy options.

Additionally, participants may be invited to review and provide feedback on the study design of heart failure trials under development, helping to ensure alignment with patient needs. Their input can identify potential procedure challenges and enhance the clarity of study materials, improving overall patient engagement. A follow-up call with a research physician will provide the opportunity to discuss any issues identified in the clinical baseline assessment and allow the participant to ask any additional questions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 45 to 80 years (inclusive) at the date of signing the informed consent.
2. Diagnosed with heart failure.
3. Able and willing to provide informed consent to participate.

Exclusion Criteria:

1. Diagnostic test results positive for:

   1. HIV-1 or HIV-2 infection
   2. Hepatitis B or Hepatitis C infection
2. Mental incapacity, language barriers or unwillingness to comply with the requirements of the protocol, which may preclude adequate understanding or cooperation during the study as judged by the Investigator.
3. Any condition judged by the Investigator to pose an undue risk while participating in the trial
4. Diagnostic results which are inconsistent with heart failure with mildly reduced or preserved ejection fraction as judged by the Investigator.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General public who meet the inclusion/exclusion criteria
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2027-01-21 (Estimated); Study Completion 2027-02-21 (Estimated)

PRIMARY OUTCOMES:
To generate high quality ECG data to establish an ECG library for the development of an ECG tool to monitor disease progression. | 18 months
  After providing informed consent, participants will then undergo a series of clinical assessments, and the participants' ECGs will be used to contribute to establishing an ECG library for future heart disease research.

SECONDARY OUTCOMES:
To gather patient perspectives on the current standard of care heart failure management and procedures. • To gather patient perspectives on preferences related to undergoing clinical diagnostics with the aim of improving the design of a disease monitor | 18 months
  Patients' perspectives on the current standard of care clinical procedures will be gathered. Patient preferences will be gathered in relation to factors around routine clinical investigations for heart failure to better design a disease monitoring tool to include clinical and patient preferences. Also, the patients may be updated on the latest therapy options.

OTHER OUTCOMES:
To gather participant feedback on the design of future heart failure trials. | 18 months
  Participants may be invited to review and provide feedback on the study design of heart failure trials under development, helping to ensure alignment with patient needs. Their input can identify potential procedure challenges and enhance the clarity of study materials, improving overall patient engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Richmond Pharmacology
Locations (1):
- Richmond Pharmacology, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Study publication when completed

REFERENCES:
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A. Corrigendum to: 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC) With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2021 Dec 21;42(48):4901. doi: 10.1093/eurheartj/ehab670. No abstract available. PMID 34649282
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992